CLINICAL TRIAL: NCT01968564
Title: Clinical Translation of Curcumin Therapy to Treat Arterial Aging
Brief Title: Oral Curcumin Supplementation in Middle-Aged and Older Adults Improves Vascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B6398
Record Dates: First submitted 2013-10-19; First posted 2013-10-24 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Vascular Aging
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High-dose curcumin pill (Experimental)
  Interventions: Drug: High-dose curcumin pill
- Low-dose curcumin pill (Experimental)
  Interventions: Drug: Low-dose curcumin pill
- Placebo pill (Placebo Comparator)
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Placebo pill — sugar and other inert substances
  Arms: Placebo pill
Drug: High-dose curcumin pill — 2000mg curcumin pill/day
  Arms: High-dose curcumin pill
Drug: Low-dose curcumin pill — 500mg curcumin pill/day
  Arms: Low-dose curcumin pill

SUMMARY:
The proposed study will assess the ability of curcumin, the active ingredient in the Indian spice tumeric, to improve the function of arteries with age. Overall, the proposed research project has the long-term potential to influence clinical practice guidelines by establishing a novel, easy to deliver, cost-effective therapy for treating age-associated arterial dysfunction and reducing the risk of cardiovascular disease with age.

ELIGIBILITY:
Inclusion Criteria:

* women must be postmenopausal
* body mass index (BMI) <40 kg/m2
* weight stable in the prior 3 months
* absence of clinical disease as determined by medical history, physical examination, blood and urine chemistries, ankle-brachial index, and a graded exercise stress test with monitoring of blood pressure and 12-lead ECG

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Arterial Stiffness | 12 weeks
  Arterial pulse wave velocity
Nitric-oxide mediated endothelium-dependent dilation | 12 weeks
  flow-mediated dilation and forearm blood flow responses to acetylcholine in the presence and absence of N'-monomethyl-L-arginine

SECONDARY OUTCOMES:
Systemic oxidative stress and inflammation | 12 weeks
  circulating markers of oxidative stress and inflammation
Endothelial cell oxidative stress and inflammation | 12 weeks
  inflammatory and oxidative stress markers in biopsied vascular and arterial endothelial cells

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Santos-Parker, MS, Study Director — University of Colorado, Boulder; Douglas Seals, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Clinical Translational Research Center, Boulder, Colorado, United States

REFERENCES:
- See also: Link Text: Description of our Research and Laboratory — http://www.colorado.edu/intphys/research/cardiovascular.html